CLINICAL TRIAL: NCT05152953
Title: Preparing for Pharmacy-based Delivery of Long-acting Injectable Antiretroviral Therapy (LAI-ART)
Status: Completed | Type: Observational
Sponsor: University of California, San Francisco (Other)
Collaborators: ViiV Healthcare (Industry); Texas A&M University (Other); Auburn University (Other); Nova Southeastern University (Other)
Responsible Party: Sponsor
Other Study IDs: 2179
Record Dates: First submitted 2021-11-29; First posted 2021-12-10 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Hiv
Keywords: pharmacy; implementation science; cabotegravir; rilpivirine; antiretroviral therapy
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Persons with HIV: Persons with HIV who are currently taking antiretroviral therapy who reside in the study's target geographical areas.
- Pharmacy staff members: Pharmacists, pharmacy technicians, pharmacy managers, or clerks employed at a community pharmacy who would potentially be involved in program development, scheduling, financial aspects, planning or administration of long-acting injectable antiretroviral therapy in the pharmacy.
- Clinic staff members: Physicians, clinic managers, nurses, medical assistants, social work staff or case managers, therapists, and other clinic personnel who are involved or would potentially be involved in any aspect of long-acting antiretrovirals in the clinic facility including financial aspects, planning, scheduling patients, educating patients, ordering medication, or administering medications.

SUMMARY:
BACKGROUND: Long-acting injectable antiretroviral therapy (LAI-ART) is poised to revolutionize HIV treatment and prevention. Community pharmacies could serve as another place for people with HIV to get their ART injections. However, pharmacist and healthcare practitioner attitudes towards pharmacist administration of LAI-ART are understudied. Financial and human resources, pharmacist training, or changes in workflow have not been outlined. Little is known about whether patients will accept ART injections given in pharmacies.

OBJECTIVE: The purpose of this project is to address the above knowledge gaps. The information generated can assist in the development of tools that can help scale community pharmacy-based delivery of LAI-ART.

METHODS: Using a mixed-methods approach to better understand the pre-implementation environment, the study will employ electronic surveys and will administer semi-structured interviews via telephone for three key stakeholder groups: HIV clinic staff members, community pharmacists, and persons with HIV. Surveys will assess the appropriateness, acceptability, and feasibility of LAI-ART administration in community pharmacies. A semi-structured interview guide has been developed using constructs from the Consolidated Framework for Implementation Research (CFIR). Comparisons between and across stakeholder groups will be performed, looking for common themes as well as discrepancies.

DETAILED DESCRIPTION:
The objective of this study is to facilitate the future delivery of long-acting injectable antiretroviral therapy in community pharmacies by developing an in-depth understanding of attitudes, barriers, and facilitators for implementing this intervention. The mixed-methods approach will incorporate three quantitative implementation outcome measures (Acceptability of Intervention Measure, Intervention Appropriateness Measure, and Feasibility of Intervention Measure) and semi-structured qualitative individual interviews which will be analyzed for relevant themes. This would be considered pure implementation research of the pre-implementation stage of LAI-ART administration in community pharmacies. Participants will be purposively sampled from four different geographical sites (San Francisco Bay Area, Corpus Christi Texas Area, Montgomery Alabama Area, and Miami/Hollywood Area) and over three different key stakeholder groups (pharmacists, patients, clinic staff) to obtain a variety of experiences, attitudes, and opinions. Most participants will have a single study visit which consists of their interview. A small proportion of pharmacists will have a second study visit for a follow up interview and questionnaire if their pharmacies have implemented a program to administer LAI-ART or are close to launching one.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or over
* Access to telephone (at minimum), access to internet/email preferred

Pharmacy staff members must meet the following additional criteria:

* Currently employed at a community (retail, independent, specialty, chain) or outpatient health system pharmacy.
* Self-reported likelihood or potential to be involved with some aspect (e.g. billing, scheduling, administering, advertising, training) of implementing long-acting injectable antiretroviral therapy in pharmacies.

Patients (persons with HIV) must meet the following additional criteria:

* Self-reported diagnosis of HIV, currently taking antiretroviral therapy (LAI-ART or oral or other)
* Self-reported undetectable HIV-1 viral load (Note: if potential participant does not know they will be encouraged to contact their health care provider to ask)
* Access to telephone

Clinic staff must meet the following additional criteria:

* Currently employed in a clinic practice where HIV-positive patients comprise > 10% of clinic population
* Self-reported likelihood or potential to be involved with some aspect (e.g. billing, scheduling, administering, advertising, training, referring patients to other clinics) of implementing long-acting injectable antiretroviral therapy in their own clinic setting.

Exclusion Criteria:

* Pharmacy staff with no forseeable involvement in implementation of a long-acting injectable antiretroviral therapy administration program.
* Patients/persons who are not diagnosed with HIV, who are candidates for long-acting cabotegravir as HIV pre-exposure prophylaxis.
* Clinic staff members with no current or forseeable involvement in supporting patients to receive long-acting injectable antiretroviral therapies.
* Persons who do not speak English to a degree that would allow full comprehension of and participation in the study.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients/persons with HIV will be recruited from local HIV clinics in the San Francisco Bay Area, Corpus Christy Texas Area, Montgomery/Opelika Alabama Area, and Miami/Hollywood Florida Areas.
  Clinic Staff Members will be recruited from HIV local clinics in the San Francisco Bay Area, Corpus Christy Texas Area, Montgomery/Opelika Alabama Area, and Miami/Hollywood Florida Areas.
  Pharmacy Staff Members will be recruited from community pharmacies serving persons with HIV that are physically located in the San Francisco Bay Area, Corpus Christy Texas Area, Montgomery/Opelika Alabama Area, and Miami/Hollywood Florida Areas.
Sampling Method: Non-Probability Sample
Enrollment: 63 (Actual)
Dates: Start 2022-06-08 (Actual); Primary Completion 2023-11-15 (Actual); Study Completion 2023-11-15 (Actual)

PRIMARY OUTCOMES:
Acceptability of intervention measure (AIM) | Baseline
  a 5-point Likert scale of agreement (1= Completely disagree, 2 = Disagree, 3 = Neither agree nor disagree, 4 = Agree, 5 = Completely agree). No items are reverse coded. Higher scores indicate greater acceptability for LAI-ART in pharmacies.
Intervention appropriateness measure (IAM) | Baseline
  a 5-point Likert scale of agreement (1= Completely disagree, 2 = Disagree, 3 = Neither agree nor disagree, 4 = Agree, 5 = Completely agree). No items are reverse coded. Higher scores indicate greater perceived appropriateness for LAI-ART in pharmacies.
Feasibility of intervention measure (FIM) | Baseline
  a 5-point Likert scale of agreement (1= Completely disagree, 2 = Disagree, 3 = Neither agree nor disagree, 4 = Agree, 5 = Completely agree). No items are reverse coded. Higher scores indicate greater perceived feasibility for LAI-ART in pharmacies.
Interview | Baseline
  Semi-structured interviews will be conducted, audio-recorded, and transcribed. Themes derived from these semi-structured individual interviews will be organized via the Consolidated Framework for Implementation Research (CFIR) and compared across the three key stakeholder groups (persons with HIV, pharmacy staff, and clinic staff).
  * Characteristics of the intervention
  * Inner setting
  * Outer setting
  * Individuals involved
  * Implementation process

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Cocohoba, PharmD, Principal Investigator — University of California San Francisco School of Pharmacy
Locations (4):
- United States (4):
  - Auburn University Harrison School of Pharmacy, Auburn, Alabama
  - University of California San Francisco School of Pharmacy, San Francisco, California
  - Nova Southeastern University College of Pharmacy, Fort Lauderdale, Florida
  - Texas A&M Irma Lerma Rangel College of Pharmacy, Kingsville, Texas

IPD SHARING:
Plan to Share IPD: Yes
De-identified data from baseline surveys and redacted interview transcripts will be made available for collaborative research
Supporting Information: Study Protocol, SAP
Time Frame: Data available upon request 6 months after initial study publication.
Access Criteria: Principal investigator will review data requests on an individual basis.